CLINICAL TRIAL: NCT01749566
Title: Exploring HIV Entry Blockade as a Pre-exposure Prophylaxis Strategy in Women
Acronym: MVC-PREP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Anandi Sheth, Assistant Professor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00059752; KL2TR000455 (NIH); ACTSIKL22012 (Other: Other)
Record Dates: First submitted 2012-11-09; First posted 2012-12-13 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: HIV
Keywords: HIV/AIDS, preexposure prophylaxis, women's health
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (standard maraviroc dosing) (Active Comparator): maraviroc 300mg po bid x 7 days
  Interventions: Drug: maraviroc
- Group B (reduced maraviroc dosing) (Active Comparator): maraviroc 300mg po daily x 7 days
  Interventions: Drug: maraviroc
- Group C (no drug) (No Intervention): No additional drug

INTERVENTIONS:
Drug: maraviroc — Maraviroc administered at standard (300mg po bid) or reduced (300mg po daily) dosing
  Other Names: Selzentry
  Arms: Group A (standard maraviroc dosing); Group B (reduced maraviroc dosing)

SUMMARY:
Pre-exposure prophylaxis (PrEP) is an HIV prevention strategy in which HIV medicines are used by a person before they are exposed to HIV in order to decrease his or her chance of getting infected. In this study, we will investigate a new PrEP strategy in women using a drug called maraviroc, a medicine used in the treatment of HIV infection called a CCR5 antagonist. We hypothesize that maraviroc could be a particularly good drug for PrEP because it achieves high concentrations in the genital tract in women and decreases the number of HIV-susceptible cells in the genital tract, and thus could potentially be dosed in more favorable ways than the current PrEP drugs.

In order to further evaluate this PrEP strategy, we plan to measure the amount of maraviroc in the blood and genital tract of HIV-negative healthy female volunteers before, during, and after they are given maraviroc dosed either in the standard (twice a day) or reduced (once a day) dose for 7 days compared with women who are not given maraviroc. We will also study immune cells from the blood and genital tract from these women to see if maravoric has an effect on these cells that would prevent them from becoming infected with HIV.

DETAILED DESCRIPTION:
RATIONALE Globally, over half of HIV-infected adults are women, and in the United States, 25% of all HIV/AIDS cases occur in women. Women often lack control over many available prevention measures, underscoring a critical need to enhance HIV prevention options for women. Pre-exposure prophylaxis (PrEP) is an HIV prevention strategy in which antiretroviral (ARV) drugs are used prior to potential HIV exposure to reduce the likelihood of infection. This strategy, which usually contains the drug tenofovir disoproxil fumarate (TDF), has recently shown promise, but efficacy data suggest room for improvement, particularly for women, in whom these data are conflicting. This study aims to prospectively examine ARV pharmacology and mucosal immunology in order to evaluate a novel PrEP strategy in women - blockade of HIV entry from its target cells at the mucosal surface using the CCR5 receptor antagonist maraviroc (MVC). These actions of CCR5 receptor antagonism, if validated, could lead to reduced HIV acquisition risk at more favorable dosing strategies than available for current PrEP. Knowledge of pharmacological modulation of mucosal immunity and HIV acquisition risk is fundamental to understanding, improving, and designing new PrEP strategies.

DESIGN This is a prospective, observational cohort study with an intensive pharmacokinetic component conducted in HIV-negative healthy women. Genital tract and whole blood samples will be collected before, during, and after treatment with 7 days of oral MVC, dosed at 300mg twice daily (standard) or 300mg daily (reduced) compared with no treatment (control). Genital tract and plasma MVC concentration will be measured using intensive pharmacokinetic sampling to generate concentration-time profiles. Peripheral blood mononuclear cells (PBMC) and endocervical cells harvested from whole blood and cervicovaginal lavage respectively will be analyzed for CCR5 receptor occupancy, the number of CCR5-expressing HIV target cells, and level of T cell activation.

DURATION 21 days after the first visit of the last participants. Enrollment is expected to take 12 months.

SAMPLE SIZE 30 subjects (10 subjects per study group)

POPULATION HIV-negative healthy women, age 18 years or older, with normal menses.

ELIGIBILITY:
Inclusion Criteria:

* Female sex, defined by sex at birth
* Age greater than or equal to 18 years
* Negative HIV serology at screening
* Normal menses (within 22-35 day intervals) for at least 3 cycles
* Intact uterus and cervix
* Normal chemistry and CBC panels at screening, including

  * Absolute neutrophil count (ANC) greater than 750/mm3
  * Hemoglobin greater than 10.0 g/dL
  * Platelet count greater than 100,000/mm3
  * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase less than 3 x upper limit of normal
  * Total bilirubin less than 2.5 x upper limit of normal
  * CrCl greater than or equal to 60 mL/min as estimated by the Cockcroft- Gault equation
* Negative hepatitis B surface antigen
* Willing to use condoms for the duration of the study and abstain from sexual intercourse for 48 hours before each genital tract sampling
* Able and willing to provide informed consent

Exclusion Criteria:

* Pregnancy (by clinical history or positive urine pregnancy test at screening)
* Breastfeeding
* Alcohol or substance use that, in the opinion of the study investigator, would interfere with the conduct of the study
* History of loop electrosurgical excision procedure (LEEP), conization, or cryosurgery
* Use of systemic hormonal contraception
* Orthostasis at screening, defined as systolic blood pressure decrease of at least 20 mm Hg or a diastolic blood pressure decrease of at least 10 mm Hg within three minutes of standing.
* Known history of heart or liver disease
* Known history of any medical condition that would interfere with conduct of the study, in the opinion of the study investigator
* Symptoms of active vaginal infection at the time of screening, including new ulcerative genital lesions or purulent and/or foul-smelling vaginal discharge
* Visible ulcerative genital lesions or purulent vaginal discharge during speculum pelvic examination performed at the time of screening
* Concomitant use of medications that interact with maraviroc or known allergy to maraviroc

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in female genital tract maraviroc concentration | Day 0, 7, 10-12

SECONDARY OUTCOMES:
Female genital tract HIV target cells | Day 0, 7, 10-12, 14, 21
  HIV target cell availability (CCR5+ CD4+ T lymphocytes) in the FGT compared with blood
Female genital tract T cell activation | Day 0, 7, 10-12, 14, 21
  T cell activation (HLA-DR+ CD38+ CD4+ T-lymphocytes) in the FGT compared with blood
Vaginal microbiome | Day 0, 7, 10-12, 14, 21
  Determine the effect of CCR5 receptor blockade on the vaginal microbiome in healthy women

CONTACTS AND LOCATIONS:
Overall Officials: Anandi Sheth, MD, Principal Investigator — Emory University School of Medicine, Department of Medicine, Division of Infectious Diseases
Locations (1):
- Grady Infectious Diseases Program, Atlanta, Georgia, United States